CLINICAL TRIAL: NCT00149032
Title: Treatment of Patients With Resistant Cancer/ Post Allogeneic Stem Cell Transplantation With Donor Lymphocytes Sensitized by Antigens Expressed by the Host
Brief Title: Treatment of Patients With Donor Lymphocytes Sensitized by Antigens Expressed by the Host
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 240801-HMO-CTIL
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2005-09

CONDITIONS: Hematological Malignancy; Neoplasm Metastasis
Keywords: Metastatic solid tumor
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Procedure: DLI sensitized against antigens expressed by the host.

SUMMARY:
Allogeneic stem cell transplantation is the only effective treatment to patients resistant to conventional chemotherapy. Donor lymphocytes infusion (DLI) serve as a routine treatment of choice for patients relapsing following allogeneic stem cell transplantation. The present proposal is presented for introducing the use of immune rather than naive donor lymphocytes for patients with resistant relapse and resistant to DLI. DLI primed in-vitro against tumor cells of host origin or against host alloantigens presented by parental alloantigens in one way mixed lymphocytes culture can induce much more than potent graft-vs-leukemia and graft-vs-tumor effects, while down-regulating graft-vs-host disease (GVHD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancy or metastatic solid tumor relapsing following allogeneic bone marrow or blood stem cell transplantation (alloBMT) or non-myeloablative stem cell transplantation resistant to DLI with no GVHD when taken off anti-GVHD prophylaxis.
* Patients with documented chimerism to confirm induction of host-vs-graft transplantation tolerance.

Exclusion Criteria:

* Patients not consenting to participate in the study, or minors without approved parental consent.
* Patients with other diseases or complications that may limit their life span other than their basic disease.
* Pregnant or lactating women.
* Non-compliant patients or patients with poor performance status with life expectancy, e.g. 6 weeks.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2001-08

PRIMARY OUTCOMES:
Introducing more effective graft vs leukemia and graft vs tumor effects with immune donor lymphocytes in patients relapsing following allogeneic bone marrow or blood stem cell transplantation

SECONDARY OUTCOMES:
Upregulating of anti-tumor effects while minimizing anti-host responses

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Slavin, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel